CLINICAL TRIAL: NCT02306174
Title: Cognitive Rehabilitation and Exposure-based Class for Compulsive Hoarding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kiara Timpano, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140644
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hoarding Disorder
Keywords: Hoarding
MeSH Terms: conditions — Hoarding Disorder; Hoarding | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Rehabilitation and Exposure-based Class for Compulsi (Experimental): Cognitive training is to improve thinking by learning new skills and strategies. The class begins with cognitive training to increase ability to carry out the skills learned later in treatment.
  Exposure therapy for discarding and acquiring helps to improve ability to make choices about possessions and learn to tolerate anxiety. Participants will face making difficult choices about items and potentially letting them go. Through repeated exposure to decisions about discarding and acquiring, distress about letting go or making choices about items will decrease over time.
  Interventions: Behavioral: Cognitive Rehabilitation and Exposure-based Class for Compulsive Hoarding

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation and Exposure-based Class for Compulsive Hoarding — The group sessions consists of 20 classes, each lasting approximately 90 minutes and may consist of some or all of the following:
  * A group agreement and a confidentiality contract
  * Homework assignments
  * Viewing informational videos about hoarding
  * Behavioral experiments including sorting and discarding exercises
  * Non-acquisition exposures
  This course is based on the Manual Cognitive Rehabilitation and Exposure/Sorting Therapy for Compulsive Hoarding (Ayers et al., 2014).

SUMMARY:
The purpose of this protocol is to investigate the effectiveness of a manualized, 20-week group cognitive rehabilitation (CR) and exposure therapy (ET) course for compulsive hoarding. The overarching aim is to understand whether this course will decrease the core symptoms of hoarding and associated features.

ELIGIBILITY:
Inclusion Criteria:

* Include:

  * Individuals who exhibit subclinical and clinical levels of hoarding disorder, as determined by the SCID interview conducted at the screening assessment, will be eligible to participate in the study. Individuals may also display clinically relevant symptoms of hoarding as indicated by scores on the Hoarding Rating Scale Interview (HRS-I) and/or on the Saving Inventory-Revised (SIR).
  * Comorbid mood and anxiety disorders are permitted.
  * English-speaking
  * Pregnant women

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Individuals who are over the age of 85
* Individuals with cognitive or physical impairments that would interfere with their participation (e.g., Dementia, uncorrected hearing)
* Participants who have current or past psychotic symptoms or current or past alcohol/substance abuse/dependence may also be excluded.
* Participants may also be excluded if they are currently in other forms of psychotherapy.
* Participants may be excluded if they have had a change in psychotropic medications within three months of the baseline assessment/first class.
* Participants may be excluded if hoarding is not their primary diagnosis.
* Prisoners

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Hoarding Rating Scale Interview | 22 weeks
  The Hoarding Rating scale has a total score ranging from 0 -40 with the higher score indicating higher symptoms of hoarding.
  This will be used to assess whether hoarding symptoms decrease as a result of treatment.
Clinician's Global Impression Improvement and Severity ratings | 22 weeks
  The CGI has a score range of 0-7 with the higher score indicating more severe symptoms.This will be used to assess whether hoarding symptoms decrease as a result of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kiara Timpano, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No